CLINICAL TRIAL: NCT00149981
Title: A Facilitated Access Program to Provide Everolimus (RAD) Maintenance for Patients Completing Therapy in RAD Trials in Solid Organ Transplantation
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRAD001A2401; 2004-001473-25
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Organ Transplantation
Keywords: Kidney, heart, lung, liver, pancreas
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: everolimus (RAD) — Everolimus

SUMMARY:
Facilitated access to everolimus until it is commercially available and reimbursable by appropriate parties

DETAILED DESCRIPTION:
This is a treatment protocol designed only to provide access to everolimus (RAD) for maintenance immunosuppression. The objectives are to facilitate the management of patients on maintenance immunosuppression therapy who are completing everolimus trials,

* To provide everolimus maintenance therapy through this access program and
* To collect and review safety data for up to 120 months or until the project has been discontinued whichever comes first.
* To collect and review safety data for up to 120 months or when Certican is commercially available in the given indication and reimbursed by appropriate payors or the project has been discontinued whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Male or female recipients of solid organ transplants
* Subject is currently enrolled in an everolimus (RAD) trial sponsored by Novartis
* Currently on investigational drug everolimus (RAD) therapy

Exclusion Criteria:

* Inability or unwillingness to comply with immunosuppressive regimen.
* Pregnancy.
* History of acute organ rejection within the last 3 months.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (129):
- United States (54):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Stanford, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Maywood, Illinois
  - Novartis Investigative Site, Des Moines, Iowa
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Livingston, New Jersey
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Valhalla, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Greenville, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Galveston, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Murray, Utah
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Charleston, West Virginia
  - Novartis Investigative Site, Madison, Wisconsin
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Australia (5):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Brazil (3):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (9):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Czechia (4):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Ostrava-Poruba
  - Novartis Investigative Site, Prague
- France (13):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Le Plessis-Robinson
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Monpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Etienne
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Villejuif
- Germany (6):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
- Italy (10):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Vicenza, VI
- Novartis Investigative Site, Auckland, New Zealand
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, San Juan, Puerto Rico
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Johannesburg, South Africa
- Spain (7):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- Taiwan (5):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (3):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Salford